CLINICAL TRIAL: NCT00938522
Title: PREtreatment of Cilostazol Loading in Elective Percutaneous Coronary Intervention to Decrease Adverse Events
Brief Title: Efficacy Study of Cilostazol Loading in Elective Percutaneous Coronary Intervention
Acronym: PRECEDE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: HC Gwon, MD, PhD, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-06-031
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Last update posted 2009-07-21 (Estimated); Status verified 2009-07

CONDITIONS: Angioplasty, Transluminal, Percutaneous Coronary
Keywords: Cilostazol loading; Angioplasty, Transluminal, Percutaneous Coronary
MeSH Terms: interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cilostazol loading (Experimental)
  Interventions: Drug: Cilostazol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cilostazol — Eligible patients were randomly assigned to cilostazol group or placebo group via the internet by the online randomization system. At least 12 h before the procedure, all patients received aspirin (300 mg loading if not taking before) and clopidogrel (300 mg loading dose). Patients in the cilostazol group received 200 mg of cilostazol (loading dose) 12 hours and 2 hours before the procedure, followed by 100 mg twice daily for 3 months.
  Arms: Cilostazol loading
Drug: Placebo — Eligible patients were randomly assigned to cilostazol group or placebo group via the internet by the online randomization system. At least 12 h before the procedure, all patients received aspirin (300 mg loading if not taking before) and clopidogrel (300 mg loading dose). Patients in the placebo group received 200 mg of placebo 12 hours and 2 hours before the procedure, followed by 100 mg twice daily for 3 months.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effect of cilostazol loading before planned PCI on major adverse cardiac and cerebrovascular events in patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective PCI
* Presence of coronary lesions amenable to stent

Exclusion Criteria:

* Cardiogenic shock
* Urgent PCI
* Hypersensitivity to aspirin, clopidogrel, or cilostazol
* LVEF < 30% or congestive heart failure
* Bleeding diathesis
* leukocyte count < 3,000/mm3 and/or platelet count < 100,000/mm3
* aspartate aminotransferase or alanine aminotransferase > 3 times upper normal; serum creatinine > 2.0 mg/dl
* noncardiac disease with a life expectancy < 1 year
* inability to follow the protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-12 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebrovascular events (MACCEs: composite of death, myocardial infarction, cerebrovascular event, and target vessel revascularization) | at 3 months after PCI

SECONDARY OUTCOMES:
Late loss on quantitative coronary angiography | 9 months after index PCI
% neointimal area [100 x (stent area-lumen area)/stent area] on IVUS | 9 months after index PCI
Major adverse cardiac and cerebrovascular events (MACCEs: composite of death, myocardial infarction, cerebrovascular event, and target vessel revascularization) | 12 months after index PCI

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon-Cheol Gwon, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea